CLINICAL TRIAL: NCT00096135
Title: Treatment of Late Isolated Extramedullary Relapse From Acute Lymphoblastic Leukemia (ALL) (Initial CR1≥ 18 Months)
Brief Title: Combination Chemotherapy and Radiation Therapy in Treating Patients With Acute Lymphoblastic Leukemia That Has Relapsed in the CNS or Testes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AALL02P2; COG-AALL02P2 (Other: Children's Oncology Group); NCI-2011-01623 (Other: NCI Trial Identifier)
Record Dates: First submitted 2004-11-09; First posted 2004-11-09 (Estimated); Results first posted 2015-08-06 (Estimated); Last update posted 2017-03-21 (Actual); Status verified 2017-02

CONDITIONS: Leukemia
Keywords: recurrent childhood acute lymphoblastic leukemia; B-cell childhood acute lymphoblastic leukemia; T-cell childhood acute lymphoblastic leukemia; TdT positive childhood acute lymphoblastic leukemia
MeSH Terms: conditions — Leukemia; Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Filgrastim; Granulocyte Colony-Stimulating Factor; Cyclophosphamide; Cytarabine; Daunorubicin; Dexamethasone; Calcium Dobesilate; Etoposide; etoposide phosphate; Leucovorin; Mercaptopurine; Methotrexate; pegaspargase; Hydrocortisone; Vincristine; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CNS Patients-Treatment (combination chemotherapy) (Experimental): All patients receive common induction (vincristine sulfate, dexamethasone, daunorubicin hydrochloride & intrathecal triple therapy (ITT: MTX, therapeutic hydrocortisone and cytarabine)), consolidation (cytarabine, pegaspargase, filgrastim, re-induction (vincristine, dexamethasone, daunorubicin), and intensification chemotherapy (MTX, leucovorin calcium, mercaptopurine, etoposide, cyclophosphamide & ITT.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: etoposide; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Radiation: radiation therapy
- Testicular Relapse Patients (Combination chemotherapy) (Experimental): All patients receive common induction (vincristine sulfate, dexamethasone, daunorubicin hydrochloride & intrathecal triple therapy (ITT: MTX, therapeutic hydrocortisone and cytarabine)), consolidation (cytarabine, pegaspargase, filgrastim, testicular radiation therapy, re-induction (vincristine, dexamethasone, daunorubicin), and intensification chemotherapy (MTX, leucovorin calcium, mercaptopurine, etoposide, cyclophosphamide & ITT.
  Interventions: Biological: filgrastim; Drug: cyclophosphamide; Drug: cytarabine; Drug: daunorubicin hydrochloride; Drug: dexamethasone; Drug: etoposide; Drug: leucovorin calcium; Drug: mercaptopurine; Drug: methotrexate; Drug: pegaspargase; Drug: therapeutic hydrocortisone; Drug: vincristine sulfate; Radiation: radiation therapy

INTERVENTIONS:
Biological: filgrastim — given subcutaneously (SC)
  Other Names: Granulocyte Colony-Stimulating Factor; r-metHuG-CSF; G-CSF; Neupogen; NSC 614629
Drug: cyclophosphamide — IV over 15-30 minutes
  Other Names: CYTOXAN; NSC #26271
Drug: cytarabine — IV over 3 hours twice daily
  Other Names: Cytosine arabinoside; Ara-C; Cytosar; NSC #6387
Drug: daunorubicin hydrochloride — IV over 15 minutes
  Other Names: Daunomycin; rubidomycin; Cerubidine; NSC #82151
Drug: dexamethasone — oral twice daily
  Other Names: Decadron; Hexadrol; Dexone; Dexameth; NSC #34521
Drug: etoposide — IV over 1 hour
  Other Names: VePesid; Etopophos; VP-16; NSC #141540
Drug: leucovorin calcium — rescue IV over 24 hours
  Other Names: LCV; Wellcovorin; citrovorum factor; folinic acid; NSC 03590
Drug: mercaptopurine — oral
  Other Names: 6-MP; Purinethol; 6-mercaptopurine; NSC #000755
Drug: methotrexate — intramuscularly (IM)
  Other Names: MTX; amethopterin; Trexall; NSC #000740
Drug: pegaspargase — intramuscularly (IM)
  Other Names: PEG-asparaginase; PEGLA; PEG-L-asparaginase; polyethylene glycol-L-asparaginase; Oncaspar; NSC 624239
Drug: therapeutic hydrocortisone
Drug: vincristine sulfate — given IV
  Other Names: Oncovin; VCR; LCR; NSC #67574
Radiation: radiation therapy — Patients with isolated testicular relapse will start Induction with a single dose of high-dose methotrexate (HDMTX) and will not receive either testicular or cranial radiation. Patients with isolated CNS relapse will NOT receive the initial dose of HDMTX prior to Induction, but will receive 1200 cGy of cranial radiation after completing the initial 12 months of intensive systemic chemotherapy.

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Giving combination chemotherapy together with radiation therapy may kill more cancer cells.

PURPOSE: This clinical trial is studying how well giving chemotherapy together with radiation therapy works in treating patients with acute lymphoblastic leukemia that has relapsed in the CNS and/or testes.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the efficacy of intensified systemic chemotherapy with reduced-dose CNS radiotherapy in patients with acute lymphoblastic leukemia and late isolated CNS relapse.
* Determine the efficacy of intensive systemic chemotherapy without testicular radiotherapy in patients with acute lymphoblastic leukemia and late isolated testicular relapse.
* Determine the toxicity of these regimens in these patients.

Secondary

* Determine whether bone marrow involvement is present at the time of extramedullary relapse in patients treated with these regimens.
* Correlate pretreatment minimal residual disease with outcomes in patients treated with these regimens.
* Correlate the role of host gene polymorphisms with toxicity of these regimens and incidence and outcome in these patients.
* Determine the neuropsychological sequelae associated with isolated CNS relapse and these treatment regimens in these patients.

OUTLINE: This is a pilot, multicenter study. All patients receive common induction, consolidation, re-induction, and intensification chemotherapy. Patients are stratified to maintenance therapy according to site of extramedullary relapse (CNS vs testicular).

* Induction therapy (weeks 1-4): Patients receive vincristine IV on days 1, 8, 15, and 22; oral dexamethasone twice daily on days 1-28; daunorubicin* IV over 15 minutes on days 1, 8, and 15; and intrathecal triple therapy** (ITT) comprising methotrexate, hydrocortisone, and cytarabine on days 1, 8, 15, and 22.

NOTE: *The total dose of anthracyclines on this study is capped at 450 mg/m2. Once this dose is reached, all subsequent doses of daunorubicin are omitted.

NOTE: **Patients with isolated testicular relapse receive ITT on day 1 only.

In addition to the above, patients with isolated testicular relapse also receive high-dose methotrexate IV continuously over 24 hours on day -14. Patients with clinical signs of disease at the end of induction undergo testicular biopsy.

Patients with CNS disease who do not achieve CNS remission after induction therapy receive additional ITT as above on days 29 and 36.

* Consolidation therapy (weeks 5-10): Patients receive high-dose cytarabine IV over 3 hours twice daily on days 1-2 and 22-23 and pegaspargase intramuscularly (IM) on days 2 and 23. Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning on days 3 and 24 and continuing until blood counts recover.

Patients with isolated testicular relapse with positive biopsy results at the end of induction undergo testicular radiotherapy once daily for a total of 12 fractions during consolidation therapy.

* Intensification I (weeks 11-22): Patients receive high-dose methotrexate with leucovorin calcium rescue IV over 24 hours on days 1, 22, 43, and 64 and oral mercaptopurine once daily on days 2-6, 23-27, 44-48, and 65-69. Patients also receive etoposide IV over 1 hour and cyclophosphamide IV over 15-30 minutes on days 8, 29, 50, and 71. Patients receive ITT* on days 15, 36, 57, and 78.

NOTE: *Patients with isolated testicular relapse receive ITT on days 36 and 78 only.

* Reinduction therapy (weeks 23-26): Patients receive vincristine IV on days 1, 8, 15, and 22; oral dexamethasone twice daily on days 1-7 and 15-21, and daunorubicin IV over 15 minutes on days 1, 8, and 15.
* Intensification II (weeks 27-50): Patients receive high-dose cytarabine IV over 3 hours twice daily on days 1-2, 43-44, 85-86, and 127-128; pegaspargase IM on days 2, 44, 86, and 128; ITT* on days 22, 64, 106, and 148; high-dose methotrexate IV continuously over 24 hours on days 29, 71, 113, and 155; oral mercaptopurine on days 30-34, 72-76, 114-118, and 156-160; and etoposide IV over 1 hour and cyclophosphamide IV over 15-30 minutes on days 36, 78, 120, and 162. Patients also receive G-CSF SC beginning on days 3, 45, 87, and 129 and continuing until blood counts recover.

NOTE: *Patients with isolated testicular relapse receive ITT on days 22 and 106 only.

* Chemotherapy and radiotherapy (weeks 51-54): Patients receive oral dexamethasone twice daily on days 1-7 and 15-21, vincristine IV on days 1, 8, and 15, and pegaspargase IM on days 1 and 15.

Patients with isolated CNS relapse also undergo cranial radiotherapy once daily, 5 days a week, for a total of 12 fractions.

* Maintenance therapy for isolated CNS relapse: (weeks 55-104): Patients receive dexamethasone PO orIV twice daily on days 1-5; oral mercaptopurine once daily on days 1-42; methotrexate IM on days 1, 8, 15, 22, 29, and 36; and vincristine IV and cyclophosphamide IV over 1 hour on days 43, 50, 57, and 64. Treatment repeats every 10 weeks for 5 courses.
* Maintenance therapy for isolated testicular relapse:

  * (Weeks 55-74): Patients receive ITT on day 1 and dexamethasone, mercaptopurine, methotrexate, vincristine, and cyclophosphamide as in maintenance therapy for isolated CNS relapse. Treatment repeats every 10 weeks for 2 courses.
  * (Weeks 75-106): Patients receive vincristine IV on day 1; dexamethasone orally or IV on days 1-5; oral mercaptopurine on days 1-28; and methotrexate IM on days 1, 8, 15, and 22. Treatment repeats every 28 days for 8 courses. Patients also receive ITT on day 1 every 12 weeks for 3 doses.

Patients with combined testicular and CNS relapse receive high-dose methotrexate IV continuously over 24 hours on day -14 in addition to the same chemotherapy and radiotherapy administered during the induction, consolidation, intensification I, reinduction, intensification II, and maintenance phases of therapy as isolated CNS relapse patients.

All patients undergo neuropsychological assessment within 3 months after completion of induction therapy (before cranial radiotherapy) and at 2 years after completion of treatment.

Patients are followed for survival.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute lymphoblastic leukemia (ALL)

  * B-precursor lineage (T-precursor lineage closed to accrual as of 05/20/10)
  * In first bone marrow remission (M1 by morphology) AND duration of first complete remission ≥ 18 months from time of initial diagnosis
* First isolated CNS and/or testicular relapse

  * Isolated CNS relapse, as defined by 1 of the following:

    * WBC ≥ 5/mm^3 in cerebrospinal fluid (CSF) with blasts present on cytospin
    * Any number of WBC in CSF with immunophenotypic proof of leukemic relapse, defined by the following:

      * Identifiable blasts AND 1 of the following:

        * B-lineage (TdT OR CD-10-positive on 2 consecutive CSF samples obtained 4 weeks apart)
        * T-lineage (TdT AND CD-7 OR TdT positivity alone on 2 consecutive CSF samples obtained 4 weeks apart) (Closed to accrual as of 05/20/10)
  * Isolated testicular relapse, defined as biopsy proven testicular involvement
* No Down syndrome
* No T-cell ALL or T-cell non-Hodgkin lymphoma
* No known optic nerve and/or retinal involvement

PATIENT CHARACTERISTICS:

Age

* 18 months to 29 years at relapse

Performance status

* Karnofsky 30-100% (for patients > 16 years of age) OR
* Lansky 30-100% (for patients ≤ 16 years of age)

Life expectancy

* Not specified

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Creatinine adjusted according to age as follows:

  * No greater than 0.4 mg/dL (≤ 5 months)
  * No greater than 0.5 mg/dL (6 months -11 months)
  * No greater than 0.6 mg/dL (1 year-23 months)
  * No greater than 0.8 mg/dL (2 years-5 years)
  * No greater than 1.0 mg/dL (6 years-9 years)
  * No greater than 1.2 mg/dL (10 years-12 years)
  * No greater than 1.4 mg/dL (13 years and over [female])
  * No greater than 1.5 mg/dL (13 years to 15 years [male])
  * No greater than 1.7 mg/dL (16 years and over [male]) OR
* Creatinine clearance or radioisotope glomerular filtration rate at least 70 mL/min

Cardiovascular

* Shortening fraction ≥ 27% by echocardiogram OR
* Ejection fraction ≥ 50% by MUGA

Other

* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior bone marrow transplantation

Chemotherapy

* Prior total anthracycline dosage ≤ 360 mg/m^2

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Other

* No prior systemic therapy for concurrent extramedullary relapse

Ages: 18 Months to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 168 (Actual)
Dates: Start 2004-11; Primary Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Julio C. Barredo, MD, Study Chair — University of Miami Miller School of Medicine-Sylvester Cancer Center; Caroline A. Hastings, MD, Study Chair — UCSF Benioff Children's Hospital Oakland
Locations (153):
- United States (135):
  - UAB Comprehensive Cancer Center, Birmingham, Alabama
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Arizona Cancer Center at University of Arizona Health Sciences Center, Tucson, Arizona
  - Arkansas Cancer Research Center at University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Southern California Permanente Medical Group, Downey, California
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Loma Linda University Cancer Institute at Loma Linda University Medical Center, Loma Linda, California
  - Jonathan Jaques Children's Cancer Center at Miller Children's Hospital, Long Beach, California
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Jonsson Comprehensive Cancer Center at UCLA, Los Angeles, California
  - Children's Hospital Central California, Madera, California
  - Children's Hospital and Research Center Oakland, Oakland, California
  - Children's Hospital of Orange County, Orange, California
  - Lucile Packard Children's Hospital at Stanford University Medical Center, Palo Alto, California
  - Sutter Cancer Center, Sacramento, California
  - Kaiser Permanente Medical Center - Oakland, Sacramento, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Children's Hospital Center for Cancer and Blood Disorders, Aurora, Colorado
  - Presbyterian - St. Luke's Medical Center, Denver, Colorado
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Broward General Medical Center Cancer Center, Fort Lauderdale, Florida
  - Lee Cancer Care of Lee Memorial Health System, Fort Myers, Florida
  - University of Florida Shands Cancer Center, Gainesville, Florida
  - Memorial Cancer Institute at Memorial Regional Hospital, Hollywood, Florida
  - Nemours Children's Clinic, Jacksonville, Florida
  - University of Miami Sylvester Comprehensive Cancer Center - Miami, Miami, Florida
  - Miami Children's Hospital, Miami, Florida
  - Baptist-South Miami Regional Cancer Program, Miami, Florida
  - Florida Hospital Cancer Institute at Florida Hospital Orlando, Orlando, Florida
  - M.D. Anderson Cancer Center at Orlando, Orlando, Florida
  - Nemours Children's Clinic - Orlando, Orlando, Florida
  - Sacred Heart Cancer Center at Sacred Heart Hospital, Pensacola, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - St. Joseph's Cancer Institute at St. Joseph's Hospital, Tampa, Florida
  - Kaplan Cancer Center at St. Mary's Medical Center, West Palm Beach, Florida
  - AFLAC Cancer Center and Blood Disorders Service of Children's Healthcare of Atlanta - Egleston Campus, Atlanta, Georgia
  - Cancer Research Center of Hawaii, Honolulu, Hawaii
  - Mountain States Tumor Institute at St. Luke's Regional Medical Center, Boise, Idaho
  - University of Illinois Cancer Center, Chicago, Illinois
  - Cardinal Bernardin Cancer Center at Loyola University Medical Center, Maywood, Illinois
  - Keyser Family Cancer Center at Advocate Hope Children's Hospital, Oak Lawn, Illinois
  - Advocate Lutheran General Cancer Care Center, Park Ridge, Illinois
  - Simmons Cooper Cancer Institute, Springfield, Illinois
  - Indiana University Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - St. Vincent Indianapolis Hospital, Indianapolis, Indiana
  - Blank Children's Hospital, Des Moines, Iowa
  - Holden Comprehensive Cancer Center at University of Iowa, Iowa City, Iowa
  - Kansas Masonic Cancer Research Institute at the University of Kansas Medical Center, Kansas City, Kansas
  - Lucille P. Markey Cancer Center at University of Kentucky, Lexington, Kentucky
  - Kosair Children's Hospital, Louisville, Kentucky
  - CancerCare of Maine at Eastern Maine Medical Center, Bangor, Maine
  - Alvin and Lois Lapidus Cancer Institute at Sinai Hospital, Baltimore, Maryland
  - Floating Hospital for Children at Tufts - New England Medical Center, Boston, Massachusetts
  - C.S. Mott Children's Hospital at University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Butterworth Hospital at Spectrum Health, Grand Rapids, Michigan
  - Van Elslander Cancer Center at St. John Hospital and Medical Center, Grosse Pointe Woods, Michigan
  - CCOP - Kalamazoo, Kalamazoo, Michigan
  - Breslin Cancer Center at Ingham Regional Medical Center, Lansing, Michigan
  - Children's Hospitals and Clinics of Minnesota - Minneapolis, Minneapolis, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - University of Mississippi Cancer Clinic, Jackson, Mississippi
  - Ellis Fischel Cancer Center at University of Missouri - Columbia, Columbia, Missouri
  - Children's Mercy Hospital, Kansas City, Missouri
  - CCOP - Nevada Cancer Research Foundation, Las Vegas, Nevada
  - Norris Cotton Cancer Center at Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Hackensack University Medical Center Cancer Center, Hackensack, New Jersey
  - Overlook Hospital, Morristown, New Jersey
  - Saint Peter's University Hospital, New Brunswick, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - St. Joseph's Hospital and Medical Center, Paterson, New Jersey
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Brooklyn Hospital Center, Brooklyn, New York
  - Maimonides Cancer Center at Maimonides Medical Center, Brooklyn, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Winthrop University Hospital, Mineola, New York
  - Schneider Children's Hospital, New Hyde Park, New York
  - NYU Cancer Institute at New York University Medical Center, New York, New York
  - Herbert Irving Comprehensive Cancer Center at Columbia University Medical Center, New York, New York
  - James P. Wilmot Cancer Center at University of Rochester Medical Center, Rochester, New York
  - Stony Brook University Cancer Center, Stony Brook, New York
  - SUNY Upstate Medical University Hospital, Syracuse, New York
  - Albert Einstein Cancer Center at Albert Einstein College of Medicine, The Bronx, New York
  - New York Medical College, Valhalla, New York
  - Blumenthal Cancer Center at Carolinas Medical Center, Charlotte, North Carolina
  - Presbyterian Cancer Center at Presbyterian Hospital, Charlotte, North Carolina
  - Duke Comprehensive Cancer Center, Durham, North Carolina
  - Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina
  - CCOP - MeritCare Hospital, Fargo, North Dakota
  - Akron Children's Hospital, Akron, Ohio
  - Rainbow Babies and Children's Hospital, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - Dayton Children's - Dayton, Dayton, Ohio
  - Medical University of Ohio Cancer Center, Toledo, Ohio
  - Tod Children's Hospital, Youngstown, Ohio
  - Oklahoma University Cancer Institute, Oklahoma City, Oklahoma
  - Legacy Emanuel Hospital and Health Center and Children's Hospital, Portland, Oregon
  - Knight Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Lehigh Valley Hospital - Muhlenberg, Bethlehem, Pennsylvania
  - Geisinger Cancer Institute at Geisinger Health, Danville, Pennsylvania
  - Penn State Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - St. Christopher's Hospital for Children, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - Rhode Island Hospital Comprehensive Cancer Center, Providence, Rhode Island
  - Hollings Cancer Center at Medical University of South Carolina, Charleston, South Carolina
  - Greenville Hospital Cancer Center, Greenville, South Carolina
  - Sanford Cancer Center at Sanford USD Medical Center, Sioux Falls, South Dakota
  - T.C. Thompson Children's Hospital, Chattanooga, Tennessee
  - East Tennessee Children's Hospital, Knoxville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Texas Tech University Health Sciences Center School of Medicine - Amarillo, Amarillo, Texas
  - Driscoll Children's Hospital, Corpus Christi, Texas
  - Medical City Dallas Hospital, Dallas, Texas
  - Simmons Comprehensive Cancer Center at University of Texas Southwestern Medical Center - Dallas, Dallas, Texas
  - Cook Children's Medical Center - Fort Worth, Fort Worth, Texas
  - Baylor University Medical Center - Houston, Houston, Texas
  - University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Methodist Children's Hospital of South Texas, San Antonio, Texas
  - Primary Children's Medical Center, Salt Lake City, Utah
  - Fletcher Allen Health Care - University Health Center Campus, Burlington, Vermont
  - Inova Fairfax Hospital, Falls Church, Virginia
  - Carilion Medical Center for Children at Roanoke Community Hospital, Roanoke, Virginia
  - Providence Cancer Center at Sacred Heart Medical Center, Spokane, Washington
  - West Virginia University Health Sciences Center - Charleston, Charleston, West Virginia
  - Mary Babb Randolph Cancer Center at West Virginia University Hospitals, Morgantown, West Virginia
  - St. Vincent Hospital Regional Cancer Center, Green Bay, Wisconsin
  - Gundersen Lutheran Center for Cancer and Blood, La Crosse, Wisconsin
  - Marshfield Clinic - Marshfield Center, Marshfield, Wisconsin
  - Midwest Children's Cancer Center at Children's Hospital of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Hospital for Children, Perth, Western Australia, Australia
- Canada (12):
  - University of Alberta Hospital, Edmonton, Alberta
  - Children's & Women's Hospital of British Columbia, Vancouver, British Columbia
  - CancerCare Manitoba, Winnipeg, Manitoba
  - Janeway Children's Health and Rehabilitation Centre, St. John's, Newfoundland and Labrador
  - IWK Health Centre, Halifax, Nova Scotia
  - McMaster Children's Hospital at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - Hopital Sainte Justine, Montreal, Quebec
  - Allan Blair Cancer Centre at Pasqua Hospital, Regina, Saskatchewan
  - Saskatoon Cancer Centre at the University of Saskatchewan, Saskatoon, Saskatchewan
  - Centre Hospitalier Universitaire de Quebec, Québec
- New Zealand (2):
  - Starship Children's Health, Auckland
  - Christchurch Hospital, Christchurch
- Switzerland (3):
  - Swiss Pediatric Oncology Group Bern, Bern
  - Swiss Pediatric Oncology Group Geneva, Geneva
  - Swiss Pediatric Oncology Group Lausanne, Lausanne

RESULTS

PARTICIPANT FLOW:
Groups:
- CNS Patients - Treatment (Combination Chemotherapy): All patients receive common induction (vincristine sulfate, dexamethasone, daunorubicin hydrochloride & intrathecal triple therapy (ITT: methotrexate, therapeutic hydrocortisone and cytarabine)), consolidation (cytarabine, pegaspargase, filgrastim, re-induction (vincristine, dexamethasone, daunorubicin), and intensification chemotherapy (methotrexate, leucovorin calcium, mercaptopurine, etoposide, cyclophosphamide & ITT.
- Testicular Relapse Patients (Combination Chemotherapy): All patients receive common induction (vincristine sulfate, dexamethasone, daunorubicin hydrochloride & intrathecal triple therapy (ITT: methotrexate, therapeutic hydrocortisone and cytarabine)), consolidation (cytarabine, pegaspargase, filgrastim, testicular radiation therapy, re-induction (vincristine, dexamethasone, daunorubicin), and intensification chemotherapy (methotrexate, leucovorin calcium, mercaptopurine, etoposide, cyclophosphamide & ITT.
Period: Overall Study
Arm/Group | CNS Patients - Treatment (Combination Chemotherapy) | Testicular Relapse Patients (Combination Chemotherapy)
Started | 126 | 42
Completed | 63 | 27
Not Completed | 63 | 15
Not completed — Physician Decision | 20 | 4
Not completed — Refusal of further protocol therapy | 4 | 1
Not completed — Progressive disease, Marrow,CNS, Relapse | 22 | 7
Not completed — Other, specify | 15 | 3
Not completed — Ineligible | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CNS Patients - Treatment (Combination Chemotherapy) | Testicular Relapse Patients (Combination Chemotherapy) | Total
Number analyzed (Participants) | 124 | 42 | 166
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 118 | 42 | 160
  Between 18 and 65 years | 6 | 0 | 6
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.2 (4.8) | 9.2 (3.2) | 8.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 0 | 36
  Male | 88 | 42 | 130
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 33 | 10 | 43
  Not Hispanic or Latino | 87 | 30 | 117
  Unknown or Not Reported | 4 | 2 | 6
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 8 | 1 | 9
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 10 | 2 | 12
  White | 91 | 33 | 124
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 15 | 6 | 21

OUTCOME MEASURES:

1. Primary Outcome: Event-free Survival
Description: Monitoring of efficacy results will be performed in comparison with historical results.
Time Frame: 3 years
Population: The CNS-treatment cohort includes 126 patients with 120 CNS pre-B, 2 CNS+ITR pre-B and 4 T-AL. The primary analysis was restricted to CNS pre-B and ITR pre-B patients, respectively. Both CNS+ITR and T-ALL patients had to be excluded from the primary analysis. That is how we came to 120 in the CNS-treatment cohort for outcome analysis.
Measure: Number; unit: percentage of participants
Arm/Group | CNS Patients - Treatment (Combination Chemotherapy) | Testicular Relapse Patients (Combination Chemotherapy)
Number analyzed (Participants) | 120 | 40
percentage of participants | 64.9 | 70

ADVERSE EVENTS:
Description: SAE field contains NCI CTCAEs submitted via expedited reporting (NCI AdEERs / CAeRs). The AE field contains grade 3 and higher CTCAEs reported on study excluding those that were reported as SAEs. The 2 ineligible patients in the CNS group are not included in the adverse event reporting.
Arm/Group | CNS Patients - Treatment (Combination Chemotherapy) | Testicular Relapse Patients (Combination Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 7/124 | 1/42
Other Adverse Events (participants affected / at risk) | 119/124 | 41/42
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNS Patients - Treatment (Combination Chemotherapy) (N=124) | Testicular Relapse Patients (Combination Chemotherapy) (N=42)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other (Cardiac disorders) | 1 (1) | 0 (0)
Death NOS (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 6 (7) | 1 (1)
Lung infection (Infections and infestations) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Fibrinogen decreased (Investigations) | 1 (1) | 0 (0)
GGT increased (Investigations) | 1 (1) | 0 (0)
INR increased (Investigations) | 1 (1) | 0 (0)
Platelet count decreased (Investigations) | 1 (1) | 0 (0)
White blood cell decreased (Investigations) | 1 (1) | 0 (0)
Acidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Adult respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CNS Patients - Treatment (Combination Chemotherapy) (N=124) | Testicular Relapse Patients (Combination Chemotherapy) (N=42)
Anemia (Blood and lymphatic system disorders) | 52 (65) | 12 (15)
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 2 (2) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 81 (86) | 27 (30)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 3 (3) | 0 (0)
Extraocular muscle paresis (Eye disorders) | 1 (1) | 0 (0)
Eye disorders - Other (Eye disorders) | 1 (1) | 1 (1)
Photophobia (Eye disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 7 (7) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Anal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 12 (12) | 5 (5)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ileus (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 15 (15) | 4 (4)
Nausea (Gastrointestinal disorders) | 7 (7) | 2 (2)
Oral pain (Gastrointestinal disorders) | 5 (5) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 4 (4) | 2 (3)
Rectal mucositis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 3 (3) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 8 (8) | 0 (0)
Death NOS (General disorders) | 0 (0) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
Fever (General disorders) | 13 (13) | 6 (6)
Flu like symptoms (General disorders) | 2 (2) | 0 (0)
General disorders and administration site conditions - Other (General disorders) | 3 (3) | 0 (0)
Multi-organ failure (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 6 (6) | 1 (1)
Sudden death NOS (General disorders) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 1 (1) | 1 (1)
Anaphylaxis (Immune system disorders) | 11 (11) | 7 (7)
Cytokine release syndrome (Immune system disorders) | 1 (1) | 1 (1)
Immune system disorders - Other (Immune system disorders) | 1 (1) | 0 (0)
Serum sickness (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Anorectal infection (Infections and infestations) | 2 (2) | 0 (0)
Arteritis infective (Infections and infestations) | 1 (1) | 0 (0)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 0 (0) | 1 (1)
Catheter related infection (Infections and infestations) | 10 (10) | 3 (3)
Enterocolitis infectious (Infections and infestations) | 6 (6) | 0 (0)
Eye infection (Infections and infestations) | 1 (1) | 0 (0)
Gum infection (Infections and infestations) | 1 (1) | 0 (0)
Infections and infestations - Other (Infections and infestations) | 82 (90) | 23 (25)
Joint infection (Infections and infestations) | 1 (1) | 0 (0)
Lung infection (Infections and infestations) | 10 (10) | 2 (2)
Meningitis (Infections and infestations) | 2 (2) | 0 (0)
Mucosal infection (Infections and infestations) | 2 (2) | 0 (0)
Otitis externa (Infections and infestations) | 4 (4) | 0 (0)
Otitis media (Infections and infestations) | 1 (1) | 0 (0)
Penile infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Salivary gland infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 4 (4) | 1 (1)
Sinusitis (Infections and infestations) | 2 (2) | 1 (1)
Skin infection (Infections and infestations) | 4 (4) | 2 (2)
Small intestine infection (Infections and infestations) | 1 (1) | 1 (1)
Upper respiratory infection (Infections and infestations) | 4 (4) | 2 (2)
Urinary tract infection (Infections and infestations) | 7 (7) | 1 (1)
Wound infection (Infections and infestations) | 3 (3) | 0 (0)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Intraoperative venous injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Activated partial thromboplastin time prolonged (Investigations) | 4 (4) | 0 (0)
Alanine aminotransferase increased (Investigations) | 64 (71) | 12 (14)
Alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 35 (35) | 4 (5)
Blood bilirubin increased (Investigations) | 7 (7) | 1 (1)
Cholesterol high (Investigations) | 2 (2) | 0 (0)
Creatinine increased (Investigations) | 2 (2) | 0 (0)
Electrocardiogram QT corrected interval prolonged (Investigations) | 0 (0) | 1 (1)
Fibrinogen decreased (Investigations) | 1 (1) | 1 (1)
GGT increased (Investigations) | 6 (6) | 0 (0)
Investigations - Other (Investigations) | 1 (1) | 0 (0)
Lipase increased (Investigations) | 9 (10) | 1 (1)
Lymphocyte count decreased (Investigations) | 3 (5) | 1 (2)
Neutrophil count decreased (Investigations) | 98 (130) | 33 (42)
Platelet count decreased (Investigations) | 73 (97) | 16 (23)
Serum amylase increased (Investigations) | 4 (4) | 0 (0)
Weight gain (Investigations) | 2 (2) | 1 (1)
White blood cell decreased (Investigations) | 63 (93) | 14 (19)
Anorexia (Metabolism and nutrition disorders) | 5 (5) | 3 (3)
Dehydration (Metabolism and nutrition disorders) | 8 (8) | 6 (6)
Glucose intolerance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycemia (Metabolism and nutrition disorders) | 9 (9) | 5 (7)
Hyperkalemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 1 (1)
Hypoalbuminemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 6 (6) | 0 (0)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 30 (35) | 9 (9)
Hypomagnesemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 12 (12) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 4 (4) | 1 (1)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Avascular necrosis (Musculoskeletal and connective tissue disorders) | 3 (3) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 6 (6) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 1 (1)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (5) | 3 (3)
Ataxia (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 1 (1) | 0 (0)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 7 (7) | 0 (0)
Memory impairment (Nervous system disorders) | 1 (1) | 0 (0)
Neuralgia (Nervous system disorders) | 1 (1) | 0 (0)
Peripheral motor neuropathy (Nervous system disorders) | 9 (9) | 2 (2)
Peripheral sensory neuropathy (Nervous system disorders) | 8 (8) | 3 (3)
Seizure (Nervous system disorders) | 2 (2) | 0 (0)
Sinus pain (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Agitation (Psychiatric disorders) | 1 (1) | 1 (1)
Anxiety (Psychiatric disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (1) | 0 (0)
Depression (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 1 (1) | 0 (0)
Personality change (Psychiatric disorders) | 2 (2) | 1 (1)
Psychosis (Psychiatric disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 0 (0)
Proteinuria (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal calculi (Renal and urinary disorders) | 0 (0) | 1 (1)
Urinary tract obstruction (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 1 (1) | 0 (0)
Penile pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Perineal pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal inflammation (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Bronchopulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 1 (1)
Pharyngeal mucositis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 (7) | 2 (2)
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Purpura (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 0 (0)
Hypotension (Vascular disorders) | 4 (4) | 3 (3)
Thromboembolic event (Vascular disorders) | 1 (1) | 3 (3)
Vascular disorders - Other (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The COG SDC reviewed the NLM notification related to ct.gov AE/SAE reporting. The information in 'Additional Description' is accurate with respect to data supplied to ct.gov.COG plans to submit data AE/SAE data consistent with the text in this field.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior sponsor approval.